CLINICAL TRIAL: NCT02432443
Title: Play and Pre-Literacy Among Young Children
Acronym: PLAY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, John Cairney, Professor, McMaster University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: INCH-0415
Record Dates: First submitted 2015-04-24; First posted 2015-05-04 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Child Development
Keywords: Motor Skills; Pre-literacy Skills; Early Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motor and pre-literacy program (Experimental): First group to receive the motor and pre-literacy program.
  Interventions: Behavioral: Motor and pre-literacy program
- Wait-list comparison (Active Comparator): Second group to receive the motor and pre-literacy program after the experimental arm has completed the program.
  Interventions: Other: Wait-list Comparison

INTERVENTIONS:
Behavioral: Motor and pre-literacy program — The program will run for 60 minutes once per week for 10 consecutive weeks and will consist of three components: direct FMS instruction, unstructured exploratory free-play, and an interactive storybook reading activity. The curriculum and teaching strategies to be used for the first two segments of our intervention have been successfully implemented in previous research to improve the motor skills of 4 year old children with autism (Bremer, Balogh, & Lloyd, 2014). Specific strategies and books were selected from an existing evidence-based curriculum (Justice & McGuinty, 2009). There will be active involvement of at least one parent in the direct instruction and reading components.
  Arms: Motor and pre-literacy program
Other: Wait-list Comparison — The participants will not participate in the motor and pre-literacy program for 10 weeks after enrollment and will continue with their normal daily life without any intervention. After the experimental arm completes the motor and pre-literacy program, the wait-list group will receive the exact same motor and pre-literacy intervention.
  Arms: Wait-list comparison

SUMMARY:
Children begin to develop fundamental motor skills (FMS), such as running and kicking, and pre-literacy skills, such as rhyming, during early childhood. These skills are very important as they lay the foundation for more complex movements and literacy skill development later in life, support overall healthy development in several areas, and help contribute to the child's readiness for school. A child with strong motor skills is well equipped to lead a life with healthy levels of physical activity, positive social interactions, positive self-perceptions, and greater cognitive and language abilities. These skills will not develop optimally on their own so it is essential to teach, challenge, and reinforce them at an early age; often this learning takes place at home prior to entering school. Most research on this topic has primarily focused on school-aged children or children with specific developmental challenges and less is known about teaching motor and pre-literacy skills to young children and giving parents the tools to practice these skills at home with their children. The aim of the present study is to examine the effect of a motor and pre-literacy program, which emphasizes parental involvement, on motor, pre-literacy, social skills, cognitive abilities, and self-competence in 3 to 4 year old children with typical development.

DETAILED DESCRIPTION:
The primary purpose of the intervention is to support the overall healthy development of children. Children will be recruited from families attending community agencies (e.g. Ontario Early Years Centres) in Hamilton. Interested parents will receive information flyers with the study team's contact information and instructions to contact the study team if they are interested in participating in the study. Interested parents will be screened for eligibility of their child. Information packages will be emailed or mailed to eligible families and will be followed-up with over the telephone in one week to obtain informed verbal consent. Baseline appointments will be booked for all eligible children. Informed written consent will be obtained at the baseline appointment before testing begins. Children will be randomized 1:1 to either the experimental or wait-list control group. Randomization will be completed using a computer algorithm. All children will be assessed pre- and post-program as well as at follow-up, 5 weeks after the completion of the program. Children in the wait-list control group will be assessed one additional time at baseline. The program will run for one hour per week for 10 consecutive weeks. Parents will be asked to complete a checklist each week indicating the number of times they practiced the activities at home. A sample size of 36 children is considered sufficient to provide 80% power to detect a medium effect size, with an alpha of 0.05. Eighteen children will be randomized to the experimental group and 18 children will be randomized to the wait-list control group.

ELIGIBILITY:
Inclusion Criteria:

* typical development

Exclusion Criteria:

* diagnosed with any developmental delay (e.g., autism, Developmental Coordination Disorder, etc.) or health conditions that may prohibit safe participation in the program (e.g., unstable heart condition).

Ages: 36 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2015-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Peabody Developmental Motor Scales-2 at 11-12 weeks | Baseline and 11-12 weeks
Change from baseline in pre-literacy skills (Phonological Awareness Literacy Screening: Preschool and Preschool Word and Print Awareness Test) at 11-12 weeks | Baseline and 11-12 weeks

SECONDARY OUTCOMES:
Change from baseline in parental engagement in motor and pre-literacy activities at 15-16 weeks | Baseline and 15-16 weeks.
Change from baseline in Peabody Developmental Motor Scales-2 at 15-16 weeks | Baseline and 15-16 weeks.
Change from baseline in Pictorial Scale of Perceived Competence and Social Acceptance for Young Children (Preschool-Kindergarten version) scale at 15-16 weeks | Baseline and 15-16 weeks.
Change from baseline in Pictorial Scale of Perceived Competence and Social Acceptance for Young Children (Preschool-Kindergarten version) scale at 11-12 weeks | Baseline and 11-12 weeks.
Change from baseline in pre-literacy skills (Phonological Awareness Literacy Screening: Preschool and Preschool Word and Print Awareness Test) at 15-16 weeks | Baseline and 15-16 weeks.
Change from baseline in Behavior Rating Inventory of Executive Function®-Preschool Version (BRIEF®-P) scale at 15-16 weeks | Baseline and 15-16 weeks.
  Parent-reported measure of executive function
Change from baseline in Behavior Rating Inventory of Executive Function®-Preschool Version (BRIEF®-P) scale at 11-12 weeks | Baseline and 11-12 weeks.
  Parent-reported measure of executive function
Change from baseline in Social Skills Improvement System (parent version) scale at 15-16 weeks | Baseline and 15-16 weeks.
  Parent-reported measure of social skills and behavioral problems
Change from baseline in Social Skills Improvement System (parent version) scale at 11-12 weeks | Baseline and 11-12 weeks.
  Parent-reported measure of social skills and behavioral problems

CONTACTS AND LOCATIONS:
Overall Officials: John Cairney, PhD, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - Boys and Girls Club of Hamilton, Hamilton, Ontario
  - McMaster Innovation Park, Hamilton, Ontario

REFERENCES:
- [Background] Boethel M. Readiness: School, Family, & Community Connections. Annual Synthesis, 2004. Southwest Educational Development Laboratory [Internet]. 2004 [cited 2015 Feb2]. Available from: http://files.eric.ed.gov/fulltext/ED484507.pdf
- [Background] Bremer E, Balogh R, Lloyd M. Effectiveness of a fundamental motor skill intervention for 4-year-old children with autism spectrum disorder: A pilot study. Autism. 2015 Nov;19(8):980-91. doi: 10.1177/1362361314557548. Epub 2014 Nov 28. PMID 25432505
- [Background] Clark JE From the beginning: a developmental perspective on movement and mobility. Quest [Internet]. 2005 [cited 2014 Dec 1]; 57(1):37-45. Available from: http://www.tandfonline.com/doi/pdf/10.1080/00336297.2005.10491841 DOI: 10.1080/00336297.2005.10491841
- [Background] Diamond A. Close interrelation of motor development and cognitive development and of the cerebellum and prefrontal cortex. Child Dev. 2000 Jan-Feb;71(1):44-56. doi: 10.1111/1467-8624.00117. PMID 10836557
- [Background] Folio MR, Fewell RR. Peabody Developmental Motor Scales--2nd Edition. 1974
- [Background] Gioia G, Espy KA, Isquith PK. Behavior Rating Inventory of Executive Function-Preschool Version (BRIEF-P). Odessa, FL: Psychological Assessment Resources; 2005.
- [Background] Gresham FM, Elliott SN. Social Skills Improvement System-Rating Scales. Minneapolis, MN: Pearson Assessments; 2008.
- [Background] Harter S, Pike R. The pictorial scale of perceived competence and social acceptance for young children. Child Dev. 1984 Dec;55(6):1969-82. PMID 6525886
- [Background] Invernizzi MA, Sullivan A, Meier JD, Swank L. Phonological Awareness Literacy Screening: Preschool Charlottesville, VA: University of Virginia; 2004.
- [Background] Isenberg JP, Quisenberry N. A position paper of the Association for Childhood Education International PLAY: Essential for all Children. Childhood Education [Internet] 2002 [cited 2015 Feb 22];79(1):33-39. Available from: http://www.tandfonline.com/doi/pdf/10.1080/00094056.2002.10522763
- [Background] Iverson JM. Developing language in a developing body: the relationship between motor development and language development. J Child Lang. 2010 Mar;37(2):229-61. doi: 10.1017/S0305000909990432. Epub 2010 Jan 25. PMID 20096145
- [Background] Justice LM, Ezell HK. Word and print awareness in 4-year old children. Child Language Teaching and Therapy [Internet] 2001 October [cited 2015 Apr 2];17(3): 207-225. Available from: http://clt.sagepub.com/content/17/3/207.full.pdf+html
- [Background] Justice LM, McGuinty AS. Read It Again-PreK!A Preschool Curriculum Supplement to Promote Language and Literacy Foundations. [Internet] 2009 [cited 2014 Oct 20]. Available from: http://arts-sciences.und.edu/communication-sciences-disorders/_files/docs/readitagain-prekmanual.pdf
- [Background] Logan SW, Robinson LE, Wilson AE, Lucas WA. Getting the fundamentals of movement: a meta-analysis of the effectiveness of motor skill interventions in children. Child Care Health Dev. 2012 May;38(3):305-15. doi: 10.1111/j.1365-2214.2011.01307.x. Epub 2011 Sep 1. PMID 21880055
- [Background] National Research Council (US) and Institute of Medicine (US) Committee on Integrating the Science of Early Childhood Development; Shonkoff JP, Phillips DA, editors. From Neurons to Neighborhoods: The Science of Early Childhood Development. Washington (DC): National Academies Press (US); 2000. Available from http://www.ncbi.nlm.nih.gov/books/NBK225557/ PMID 25077268
- [Derived] Bedard C, Bremer E, Campbell W, Cairney J. Evaluation of a Direct-Instruction Intervention to Improve Movement and Preliteracy Skills among Young Children: A Within-Subject Repeated-Measures Design. Front Pediatr. 2018 Jan 17;5:298. doi: 10.3389/fped.2017.00298. eCollection 2017. PMID 29387681
- [Derived] Bedard C, Bremer E, Campbell W, Cairney J. A Quasi-Experimental Study of a Movement and Preliteracy Program for 3- and 4-Year-Old Children. Front Pediatr. 2017 May 1;5:94. doi: 10.3389/fped.2017.00094. eCollection 2017. PMID 28507981